CLINICAL TRIAL: NCT02299440
Title: Evaluation of the Effects of Ketamine in the Acute Phase of Suicidal Ideation: a Multicenter Randomized Double-blind Trial
Brief Title: Effects of Ketamine in the Acute Phase of Suicidal Ideation
Acronym: KETIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC-N/2013/MA-01; 2014-001324-30 (EudraCT Number)
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2019-03

CONDITIONS: Suicidal Ideation
Keywords: treatment of acute suicidal ideation; ketamine; low-dose ketamine
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Patients randomized to this group will be treated via Ketamine infusion.
  Intervention: Baseline evaluation Intervention: 1st perfusion of ketamine Intervention: Follow-up between perfusions Intervention: 2nd perfusion of ketamine Intervention: Follow-up after perfusions
  Interventions: Other: Baseline evaluation; Drug: 1st perfusion of ketamine; Other: Follow-up between perfusions; Drug: 2nd perfusion of ketamine
- Placebo/Control (Placebo Comparator): Patients randomized to this group will be treated via saline solution infusion.
  Intervention: Baseline evaluation Intervention: 1st perfusion of saline Intervention: Follow-up between perfusions Intervention: 2nd perfusion of saline Intervention: Follow-up after perfusions
  Interventions: Other: Baseline evaluation; Drug: 1st perfusion of saline; Other: Follow-up between perfusions; Drug: 2nd perfusion of saline

INTERVENTIONS:
Other: Baseline evaluation — Before perfusions begin, each patient will have a baseline evaluation including the following: the Columbia Suicide Severity Rating Scale (CSSRS), the Beck Scale for Suicide Ideation (BSSI), a physical pain VAS (visual analog scale), a mental pain VAS, the Clinical Global Impressions Scale (CGI-S), Beck's Hopeless scale (BHS), the Inventory of Depressive Symptomatology for the Clinician (IDS-C30), the Patient Rated Inventory of Side Effects (PRISE), the Young Mania Rating Scale (YMRS) and the Brief Psychiatric Rating Scale (BPRS).
Drug: 1st perfusion of ketamine — A 1st perfusion of ketamine is performed: 0.5 mg/kg diluted in saline, administered over 40 minutes by intravenous (IV) pump and cardiorespiratory monitoring. (Day 0)
  Arms: Ketamine
Drug: 1st perfusion of saline — A 1st perfusion of saline is performed: the same volume of saline as in the ketamine arm, administered over 40 minutes by IV pump and cardiorespiratory monitoring. (Day 0)
  Arms: Placebo/Control
Other: Follow-up between perfusions — Patients will be re-evaluated with a selection of questionnaires at 40 minutes, 120 minutes, 4 hours, and 24 hours after the end of the first perfusion, and then again at 48 hours after the end of the first perfusion and right before the second perfusion and then again Day 3, Day 4, Week 2, Week 4 and Week 6.
Drug: 2nd perfusion of ketamine — A 2nd perfusion of ketamine is performed: 0.5 mg/kg diluted in saline, administered over 40 minutes by intravenous (IV) pump and cardiorespiratory monitoring. (Day 2)
  Arms: Ketamine
Drug: 2nd perfusion of saline — A 2nd perfusion of saline is performed: the same volume of saline as in the ketamine arm, administered over 40 minutes by IV pump and cardiorespiratory monitoring. (Day 2)
  Arms: Placebo/Control

SUMMARY:
The primary objective of this study is to assess the efficacy of ketamine versus a placebo for the short-term (at 72h, i.e. 24h after the last perfusion) relief of suicidal ideation, measured using the BSS hetero questionnaire, in patients hospitalized for suicide risk.

DETAILED DESCRIPTION:
The secondary objectives of this study are to assess:

A. The maintenance of medium-term effectiveness of ketamine on the resolution of suicidal ideation

B. The evolution of the full spectrum of suicidality under ketamine compared to placebo

C. The evolution of psychic and physical pain scores under ketamine compared to placebo

D. The evolution of Beck Hopelessness score which is a predictor of long-term suicide risk, under ketamine compared to placebo

E. The early antidepressant efficacy of ketamine in depressed, uni- or bipolar patients

F. The somatic and psychological tolerance of ketamine

G. An overall improvement in the clinical condition of the patient by the practitioner

H. Creation of a biological collection for future ancillary studies dedicated to genetic analysis (microRNA and mRNA).

I. The efficacy of ketamine versus a placebo for the short-term (at 72h, i.e. 24h after the last perfusion) relief of suicidal ideation, measured using the BSS self-report questionnaire, in patients hospitalized for suicide risk.

ELIGIBILITY:
Inclusion Criteria:

* French speaking patients freely hospitalized for prevention of suicide and who have a medium or high suicide risk score according to a MINI structured interview
* The patient is able to understand how the study is carried out and the tests performed
* The patient is deemed capable of giving his/her informed consent
* The patient has been correctly informed
* The patient must have given his/her informed and signed consent.
* The patient must be insured or beneficiary of a health insurance plan.
* Presence of suicidal ideation according to the SSI score (score > 3)
* Negative pregnancy test for women of childbearing age

Exclusion Criteria:

* The patient is participating in another interventional study
* Within the past three months, the patient has participated in another interventional study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection
* The patient is an adult under guardianship
* The patient refuses to sign the consent
* The patient is not able to understand the informed consent
* Pregnancy or breastfeeding
* History of schizophrenia or other psychotic disorders
* Presence of psychotic symptoms at initial interview
* Schizoid or schizotypic personality disorder
* Positive urine screening for illicit substances, excluding cannabis
* Substance dependence in the preceding month (excluding nicotine or caffeine)
* Concomitant treatment with electroconvulsive therapy
* Unstable somatic pathology
* Clinically significant anomalies found during clinical examination, biological test or ECG
* Non-stabilized hypertension or hypertension > 180/100
* Known or suspected contra-indication for ketamine (includes interactions): hypersensitivity to ketamine, hypertension, class IV cardiac insufficiency, history of stroke, hepatic or cutaneous porphyria, history of intracranial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
BSSI score | Day 3
  A suicidal ideation score measured using the BSS (Beck et al. 1979) in its hetero questionnaire form ≤ 3 at 24 hours after the second infusion of ketamine or placebo (yes/no). A threshold ≤ 3 separates the resolution of suicidal ideas from their persistence (Holi et al. 2005; DiazGranados et al. 2010).

SECONDARY OUTCOMES:
The occurrence of a suicide attempt or a completed suicide (yes/no) | 6 weeks
Evaluation of the full spectrum of suicidality using the CSSRS | Baseline (Day-2 to Day 0)
Evaluation of the full spectrum of suicidality using the CSSRS | Day 1
Evaluation of the full spectrum of suicidality using the CSSRS | Day 2
Evaluation of the full spectrum of suicidality using the CSSRS | Day 3
Evaluation of the full spectrum of suicidality using the CSSRS | Day 4
Evaluation of the full spectrum of suicidality using the CSSRS | Week 2
Evaluation of the full spectrum of suicidality using the CSSRS | Week 4
Evaluation of the full spectrum of suicidality using the CSSRS | Week 6
The BSSI score | Baseline (Day-2 to Day 0)
The BSSI score | 40 min after end of 1st perfusion (Day 0)
The BSSI score | 120 min after end of 1st perfusion (Day 0)
The BSSI score | 4 hours after end of 1st perfusion (Day 0)
The BSSI score | Day 1
The BSSI score | Day 2
The BSSI score | Day 4
The BSSI score | Week 2
The BSSI score | Week 4
The BSSI score | Week 6
Evaluation of physical pain using a visual analog scale of 0 to 10 following a Lickert model | Baseline (Day-2 to Day 0)
Evaluation of physical pain using a visual analog scale of 0 to 10 following a Lickert model | 40 min after end of 1st perfusion (Day 0)
Evaluation of physical pain using a visual analog scale of 0 to 10 following a Lickert model | 120 min after end of 1st perfusion (Day 0)
Evaluation of physical pain using a visual analog scale of 0 to 10 following a Lickert model | 4 hours after end of 1st perfusion (Day 0)
Evaluation of physical pain using a visual analog scale of 0 to 10 following a Lickert model | Day 1
Evaluation of physical pain using a visual analog scale of 0 to 10 following a Lickert model | Day 2
Evaluation of physical pain using a visual analog scale of 0 to 10 following a Lickert model | Day 3
Evaluation of physical pain using a visual analog scale of 0 to 10 following a Lickert model | Day 4
Evaluation of physical pain using a visual analog scale of 0 to 10 following a Lickert model | Week 2
Evaluation of physical pain using a visual analog scale of 0 to 10 following a Lickert model | Week 4
Evaluation of physical pain using a visual analog scale of 0 to 10 following a Lickert model | Week 6
Evaluation of mental pain using a visual analog scale of 0 to 10 following a Lickert model | Baseline (Day-2 to Day 0)
Evaluation of mental pain using a visual analog scale of 0 to 10 following a Lickert model | 40 min after end of 1st perfusion (Day 0)
Evaluation of mental pain using a visual analog scale of 0 to 10 following a Lickert model | 120 min after end of 1st perfusion (Day 0)
Evaluation of mental pain using a visual analog scale of 0 to 10 following a Lickert model | 4 hours after end of 1st perfusion (Day 0)
Evaluation of mental pain using a visual analog scale of 0 to 10 following a Lickert model | Day 1
Evaluation of mental pain using a visual analog scale of 0 to 10 following a Lickert model | Day 2
Evaluation of mental pain using a visual analog scale of 0 to 10 following a Lickert model | Day 3
Evaluation of mental pain using a visual analog scale of 0 to 10 following a Lickert model | Day 4
Evaluation of mental pain using a visual analog scale of 0 to 10 following a Lickert model | Week 2
Evaluation of mental pain using a visual analog scale of 0 to 10 following a Lickert model | Week 4
Evaluation of mental pain using a visual analog scale of 0 to 10 following a Lickert model | Week 6
Evaluation of despair using the Beck Hopelessness Scale | Baseline (Day-2 to Day 0)
Evaluation of despair using the Beck Hopelessness Scale | Day 1
Evaluation of despair using the Beck Hopelessness Scale | Day 2
Evaluation of despair using the Beck Hopelessness Scale | Day 3
Evaluation of despair using the Beck Hopelessness Scale | Day 4
Evaluation of despair using the Beck Hopelessness Scale | Week 2
Evaluation of despair using the Beck Hopelessness Scale | Week 4
Evaluation of despair using the Beck Hopelessness Scale | Week 6
Evaluation of depression by the clinician (IDS-C30) | Baseline (Day-2 to Day 0)
Evaluation of depression by the clinician (IDS-C30) | 4 hours after end of 1st perfusion (Day 0)
Evaluation of depression by the clinician (IDS-C30) | Day 1
Evaluation of depression by the clinician (IDS-C30) | Day 2
Evaluation of depression by the clinician (IDS-C30) | Day 3
Evaluation of depression by the clinician (IDS-C30) | Day 4
Evaluation of depression by the clinician (IDS-C30) | Week 2
Evaluation of depression by the clinician (IDS-C30) | Week 4
Evaluation of depression by the clinician (IDS-C30) | Week 6
Evaluation of somatic tolerance of ketamine using the Patient Rated Inventory of Side Effects (PRISE) throughout follow-up | Baseline (Day-2 to Day 0)
Evaluation of somatic tolerance of ketamine using the Patient Rated Inventory of Side Effects (PRISE) throughout follow-up | Day 1
Evaluation of somatic tolerance of ketamine using the Patient Rated Inventory of Side Effects (PRISE) throughout follow-up | Day 2
Evaluation of somatic tolerance of ketamine using the Patient Rated Inventory of Side Effects (PRISE) throughout follow-up | Day 3
Evaluation of somatic tolerance of ketamine using the Patient Rated Inventory of Side Effects (PRISE) throughout follow-up | Day 4
Evaluation of psychic tolerance using the Young Mania Rating Scale (YMRS) | Baseline (Day-2 to Day 0)
Evaluation of psychic tolerance using the Young Mania Rating Scale (YMRS) | Day 1
Evaluation of psychic tolerance using the Young Mania Rating Scale (YMRS) | Day 2
Evaluation of psychic tolerance using the Young Mania Rating Scale (YMRS) | Day 3
Evaluation of psychic tolerance using the Young Mania Rating Scale (YMRS) | Day 4
Evaluation of psychic tolerance using the Brief Psychiatric Rating Scale (BPRS) | Baseline (Day-2 to Day 0)
Evaluation of psychic tolerance using the Brief Psychiatric Rating Scale (BPRS) | Day 1
Evaluation of psychic tolerance using the Brief Psychiatric Rating Scale (BPRS) | Day 2
Evaluation of psychic tolerance using the Brief Psychiatric Rating Scale (BPRS) | Day 3
Evaluation of psychic tolerance using the Brief Psychiatric Rating Scale (BPRS) | Day 4
Presence/absence of abnormal monitoring values throughout the study: hypertension | 6 weeks
  Any abnormal hypertension, pulse oxymetry or cardiac frequency values observed during the study will be noted.
Presence/absence of abnormal monitoring values throughout the study: pulse oxymetry | 6 weeks
  Any abnormal hypertension, pulse oxymetry or cardiac frequency values observed during the study will be noted.
Presence/absence of abnormal monitoring values throughout the study: cardiac frequency | 6 weeks
  Any abnormal hypertension, pulse oxymetry or cardiac frequency values observed during the study will be noted.
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | Baseline (Day-2 to Day 0)
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | 40 min after end of 1st perfusion (Day 0)
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | 120 min after end of 1st perfusion (Day 0)
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | 4 hours after end of 1st perfusion (Day 0)
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | Day 1
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | Day 2
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | 120 min after end of 2nd perfusion (Day 2)
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | Day 3
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | Day 4
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | Week 2
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | Week 4
Evaluation of the improvement of the patient's clinical condition using the Clinical Global Impression scale - Improvement (CGI-I) | Week 6
The BSSI score | 24 hours after the last perfusion
  A suicidal ideation score measured using the BSS (Beck et al. 1979) in its self report questionnaire form ≤ 3 at 24 hours after the second infusion of ketamine or placebo (yes/no). This scale is validated in French (de Man, Balkou & Iglesias 1987); a threshold ≤ 3 separates the resolution of suicidal ideas from their persistence (Holi et al. 2005; DiazGranados et al. 2010)

CONTACTS AND LOCATIONS:
Overall Officials: Mocrane Abbar, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (9):
- France (9):
  - CHU de Clermont Ferrand - Hôpital Gabriel-Montpied, Clermont-Ferrand
  - CHRU de Lille - Hôpital Michel Fontan, Lille
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier
  - Clinique Les Sophoras, Nîmes
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - APHP - Hôpital Lariboisière, Paris
  - Centre Hospitalier Sainte-Anne, Paris
  - CMME Centre Hospitalier Sainte Anne, Paris
  - CHRU de Tours - Clinique Psychiatrique Universitaire, Saint-Cyr-sur-Loire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbar M, Demattei C, El-Hage W, Llorca PM, Samalin L, Demaricourt P, Gaillard R, Courtet P, Vaiva G, Gorwood P, Fabbro P, Jollant F. Ketamine for the acute treatment of severe suicidal ideation: double blind, randomised placebo controlled trial. BMJ. 2022 Feb 2;376:e067194. doi: 10.1136/bmj-2021-067194. PMID 35110300
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617